CLINICAL TRIAL: NCT05328960
Title: An Analysis of Covid-19 Effect on Patients With Colorectal Cancer - Follow-up Regarding Tumour Stage, Neoadjuvant Treatment, Delay and Long-term Survival
Brief Title: The Pandemic's Effect on Diagnosis and Treatment of Rectal Cancer
Acronym: CovidRC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor, Sahlgrenska University Hospital
Other Study IDs: CovidRC
Record Dates: First submitted 2022-04-13; First posted 2022-04-14 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed before, during or after the pandemic: Patients with rectal cancer
  Interventions: Other: Diagnosed during or not during the pandemic

INTERVENTIONS:
Other: Diagnosed during or not during the pandemic — We will create a group of patients that are diagnosed before and after the pandemic and one group diagnosed during the pandemic

SUMMARY:
Colorectal cancer is common with an annual prevalence of 6000. The majority can be cured and the five year survival rate is over 60%. In december 2019 reports came in about SARS-Cov-2, which later was named Covid-19. The World Health Organization classified it as a pandemic in March 2020. In Sweden the number of patients with Covid-19 increased mainly in the urban areas in March 2020. Care for patients with other diseases were affected and local changes from guidelines were adopted. In some regions and countries the indications for adjuvant and neoadjuvant treatment for colorectal cancer were somewhat changed. The number of patients diagnosed with colorectal cancer also decreased, as well as other types of cancer. The true effect on outcome with a delayed diagnosis remains unknown.

The aim of this study is to evaluate the effects of the Covid-19 pandemic on the diagnosis, treatment and survival of patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer diagnosis 2019-2022

Exclusion Criteria:

* No rectal cancer diagnosis 2019-2022

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are diagnosed with rectal cancer and identified in the Swedish ColoRectal Cancer Registry will be included. They will be contacted by phone and mail regarding a questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Yearly incidence of rectal cancer | 2019-2022
  The number of patients diagnosed yearly 2019, 2020, 2021 and 2022

SECONDARY OUTCOMES:
Symptoms at diagnosis | 6 months prior diagnosis
  Symptoms at diagnosis as reported by patients
Patient's delay | 12 months prior diagnosis
  Delay from symptoms until doctors appointment
Doctor's delay | 12 months prior diagnosis
  Delay from doctor's appointment until diagnosis
Treatment changes | Diagnosis and 12 months following
  Any changes from the treatment plan due to covid-19

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided